CLINICAL TRIAL: NCT04788004
Title: Long-term Recovery: Longitudinal Study of Neuro-behavioral Markers of Recovery and Precipitants of Relapse
Status: Active, not recruiting | Type: Observational
Sponsor: Virginia Polytechnic Institute and State University (Other)
Responsible Party: Principal Investigator, Jungmeen Kim-Spoon, Principal investigator, Virginia Polytechnic Institute and State University
Other Study IDs: IQRR- Longitudinal Study
Record Dates: First submitted 2021-03-03; First posted 2021-03-09 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Alcohol Use Disorder
MeSH Terms: conditions — Alcoholism

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (10):
- Cohort 1: Participants in this group started their recovery process < 1 year ago
  Interventions: Other: Online survey
- Cohort 2: Participants in this group started their recovery process 1 to <2 years ago
  Interventions: Other: Online survey
- Cohort 3: Participants in this group started their recovery process 2 to <3 years ago
  Interventions: Other: Online survey
- Cohort 4: Participants in this group started their recovery process 3 to <4 years ago
  Interventions: Other: Online survey
- Cohort 5: Participants in this group started their recovery process 4 to <5 years ago
  Interventions: Other: Online survey
- Cohort 6: Participants in this group started their recovery process 5 to <6 years ago
  Interventions: Other: Online survey
- Cohort 7: Participants in this group started their recovery process 6 to <7 years ago
  Interventions: Other: Online survey
- Cohort 8: Participants in this group started their recovery process 7 to <8 years ago
  Interventions: Other: Online survey
- Cohort 9: Participants in this group started their recovery process 8 to <9 years ago
  Interventions: Other: Online survey
- Cohort 10: Participants in this group started their recovery process 9 to <10 years ago
  Interventions: Other: Online survey

INTERVENTIONS:
Other: Online survey — There are no interventions planned for this study. This is an observational study only.

SUMMARY:
The goals of this study are to provide a scientific understanding of recovery and relapse, as well as to identify novel targets for future relapse prevention interventions.

DETAILED DESCRIPTION:
The study will characterize long-term trajectories of recovery from alcohol use including the associated changes in psychosocial functioning and relapse status. By using an accelerated longitudinal design, competing neurobehavioral decision systems (CNDS) functioning (measured using delay discounting), psychosocial functioning, and relapse will be characterized over a 12-year period for individuals in alcohol use disorder (AUD) recovery.

ELIGIBILITY:
Inclusion Criteria:

1. be ≥18 yrs old
2. meet lifetime DSM-5 AUD criteria
3. have a Recovery Initiation Date less than 10 years prior to the time of enrollment
4. be able to read independently
5. be free of legal problems that could limit participation
6. reside in the U.S.
7. anticipate continued Internet access (to ensure ongoing contact and data collection)
8. be a registrant of the International Quit and Recovery Registry (IQRR)

Exclusion Criteria:

* Minors will not be included
* Prisoners will not be included. If participants become incarcerated during this study, they will not be contacted to complete assessments during their incarceration. If the incarcerations ends during the study, they may be contacted to participate in assessments.
* Adults who are not capable of consenting on their own behalf

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Individuals in recovery from AUD who meets the study inclusion criteria will be recruited from The International Quit & Recovery Registry (IQRR) (https://quitandrecovery.org). Participants will be recruited from existing or new IQRR registrants; that is, IQRR registrants meeting the inclusion criteria (see above) will be invited to participate. Also, the recruitment of new registrants will use methods designed to reflect the heterogeneity of the recovery population.
Sampling Method: Non-Probability Sample
Enrollment: 733 (Actual)
Dates: Start 2022-09-08 (Actual); Primary Completion 2026-07-20 (Estimated); Study Completion 2026-07-20 (Estimated)

PRIMARY OUTCOMES:
CNDS functioning | Approximately every 3 months from date of baseline session through study completion, an average of 3 years
  Delay Discounting (DD) task will be administered to assesses the value of delayed reinforcers. Participants make hypothetical choices between amounts of delayed and immediate money at various delays (e.g., 1 day to 25 years)
Psychosocial Functioning- The Psychosocial Functioning Inventory (PFI) | Approximately every 3 months from date of baseline session through study completion, an average of 3 years
  The Psychosocial Functioning Inventory (PFI) will be used to measure social functioning. The social behavior sub-scale will be calculated from 10 items of the PFI and included items that assess the frequency of problematic social behavior and social interactions in the past 90 days. The psychosocial functioning scale yields a score ranging from 0-100, with higher scores indicating greater impairment.
Psychosocial Functioning- World Health Organization (WHO)-Quality of Life | Approximately every 3 months from date of baseline session through study completion, an average of 3 years
  WHO-Quality of Life brief assessment (BREF) will be used to measure the four domains of quality of life: (1) physical health; (2) psychological (3) social relationships; and (4) environment (26 items). Each item in the WHOQOL-BREF will be scored with a 5-point Likert scale (three items are reverse scored), and these scores will be used to generate raw scores for each domain, which will be then scaled 0-100, with higher scores indicating greater quality of life.
Psychosocial Functioning- Satisfaction with Life and social Functioning | Approximately every 3 months from date of baseline session through study completion, an average of 3 years
  Satisfaction with life and social functioning over the past 90 days will be assessed using 4 questions: How happy have you been (1) with life?; (2) with your living situation? and (3) with your relationships? and (4) Did you feel satisfied with leisure, social, and recreational activities? (0 = satisfied/happy; 1 = dissatisfied/unhappy)
Psychosocial Functioning- Career Engagement | Approximately every 3 months from date of baseline session through study completion, an average of 3 years
  Engagement in proactive career behaviors over time (9 items). Each item in the career engagement measure will be scored with the 5-point Likert-type scale. The average scale scores will range between 1-5 with higher score indicating greater engagement.
Psychosocial Functioning- Addiction Severity | Approximately every 3 months from date of baseline session through study completion, an average of 3 years
  The Addiction Severity Index (ASI) will be used to assess experiences of serious depression, serious anxiety or tension, and cognitive difficulty (i.e., trouble understanding, concentrating, or remembering) in the past 90 days. All items will be binary indicators, where 0 = employed or symptom not present and 1 = unemployed or symptom present. Items will be examined individually.
Alcohol Use- AUD Status and Severity | Approximately every 3 months from date of baseline session through study completion, an average of 3 years
  The Diagnostic and Statistical Manual-5 (DSM-5) AUD (last year & last 3 months) will be used to assess AUD status and severity with mild, moderate, and severe sub-classifications
Alcohol Use- Consumption | Approximately every 3 months from date of baseline session through study completion, an average of 3 years
  Timeline Follow Back-90 (TLFB-90) will be used to obtains retrospective daily estimates of alcohol consumption in the last 3 month. TLFB can generate a variety of variables that provide more precise and varied information (e.g., pattern, variability, drinking levels) about a person's drinking
Adverse Social and emotional events | Approximately every 3 months from date of baseline session through study completion, an average of 3 years
  Inventory of Drug Taking Situations (IDTS-8) will be used to assess the frequency of common relapse-inducing events (i.e., negative affect, social pressure, physical discomfort, and drinking-related variables such as temptations, urges, and alcohol cues; 8 items)

CONTACTS AND LOCATIONS:
Overall Officials: Jungmeen Kim-Spoon, PhD, Principal Investigator — Virginia Polytechnic Institute and State University; Allison Tegge, PhD, Principal Investigator — Virginia Polytechnic Institute and State University
Locations (1):
- Fralin Biomedical Research Institute at VTC, Roanoke, Virginia, United States

IPD SHARING:
Plan to Share IPD: Undecided